CLINICAL TRIAL: NCT00368043
Title: Biobehavioral Study of Recently Adopted Children
Brief Title: Endocrine and Psychological Evaluation of Adopted Children
Status: Terminated | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 060223; 06-CH-0223
Record Dates: First submitted 2006-08-23; First posted 2006-08-24 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2015-03-30

CONDITIONS: Psychosocial Adjustment
Keywords: Pituitary; Adrenal; Growth; Cortisol; Stress Response; Adoption; Thyroid Hormone; Psychosocial Adjustment; Healthy Volunteer; HV
MeSH Terms: conditions — Pituitary Diseases; Fractures, Stress

SUMMARY:
The deleterious effects of institutionalized care on the health and growth and development of children have been described. Early studies have shown that the effects of institutionalized care on a child's growth and development may not be fully reversible. The exact mechanism through which these early stresses affect bio-behavioral outcomes has yet to be determined. A likely mechanism in which environmental influences could regulate both biological and psychosocial development may be through the hypothalamic pituitary adrenal axis (HPA). Recent advances in the area of brain research have enriched our understanding of the importance of early life experiences on physical, cognitive, developmental, mental and behavioral health outcomes. Children adopted from orphanages in countries as diverse as the former Soviet Union and Guatemala provide an opportunity to learn more about the effect of deprivation on neuro-endocrine function, physical growth, and developmental outcomes, including cognitive, and behavioral measures.

This protocol proposes to study the changes of the HPA axis of the post-institutionalized adoptive child, ages 10 months to 4 years, which may help elucidate the etiology of the complex findings in this population. We will recruit 60 adopted children who experienced institutionalized care and were recently adopted by a US family and 60 controls. Our primary hypothesis is that a number of adopted children will have biochemical evidence of stress-induced activation of the HPA axis and sympathetic adrenal medullary system. HPA dysfunction will be evident by abnormal diurnal salivary cortisol levels, increased cortisol and/or catecholamine excretion in 24 hours urine measurements, and dysregulation of autonomic nervous system activity We also hypothesize that many of these responses will not normalize with time and that there will be a correlation between these responses and growth and behavioral disorders. In addition, we will examine nutritional intake and sleep patterns to determine their effect on growth and developmental outcome.

DETAILED DESCRIPTION:
The deleterious effects of institutionalized care on the health and growth and development of children have been described. Early studies have shown that the effects of institutionalized care on a child's growth and development may not be fully reversible. The exact mechanism through which these early stresses affect bio-behavioral outcomes has yet to be determined. A likely mechanism in which environmental influences could regulate both biological and psychosocial development may be through the hypothalamic pituitary adrenal axis (HPA). Recent advances in the area of brain research have enriched our understanding of the importance of early life experiences on physical, cognitive, developmental, mental and behavioral health outcomes. Children adopted from orphanages in countries as diverse as the former Soviet Union and Guatemala provide an opportunity to learn more about the effect of deprivation on neuro-endocrine function, physical growth, and developmental outcomes, including cognitive and behavioral measures.

This protocol proposes to study the changes of the HPA axis of the post-institutionalized adoptive child, ages 10 months to 4 years, which may help elucidate the etiology of the complex findings in this population. We will recruit 60 adopted children who experienced institutionalized care and were recently adopted by a US family and 60 controls. Our primary hypothesis is that a number of adopted children will have biochemical evidence of stress-induced activation of the HPA axis and sympathetic adrenal medullary system. HPA dysfunction will be evident by abnormal diurnal salivary cortisol levels, increased cortisol and/or catecholamine excretion in 24 hours urine measurements, and dysregulation of autonomic nervous system activity We also hypothesize that many of these responses will not normalize with time and that there will be a correlation between these responses and growth and behavioral disorders. In addition, we will examine nutritional intake and sleep patterns to determine their effect on growth and developmental outcome.

ELIGIBILITY:
* INCLUSION CRITERIA:

A. The patient sample will be children ages 10 months to 4 years old (pre-pubertal, Tanner I) referred to the International Adoption Center or Johns Hopkins University Medical Center for an initial evaluation within two to four weeks after they arrive from their country of origin (Eastern Europe/Russia).

A total of 60 children, ages 10 months to 6 years, will be recruited for a control group and will be frequency matched with the adopted subjects into four strata: 10 to 42 month old boys, 10 to 42 month old girls, 43 to 72 month old boys, and 43 to 72 month old girls.

The controls will be healthy children with no history of medical or psychological disorders

The controls will be healthy children with no history of medical or psychological disorders.

EXCLUSION CRITERIA:

1. Children with known documented growth hormone deficiency, and/or history of chronic illness such as renal failure, severe chronic lung disease (restrictive, obstructive) diabetes, hypothyroidism.
2. Children with known genetic or chromosomal abnormalities.
3. Children with medical conditions known to be associated with permanent developmental delay (i.e. fetal alcohol syndrome).
4. Children with chronic medication use.
5. Children with behavior problems receiving psychiatric treatment
6. Children with documented infectious diseases (AIDS, Hepatitis, etc).
7. Children with clinical signs of puberty; only children in Tanner-I pubertal stage will be allowed in the study.

Ages: 10 Months to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 38 (Actual)
Dates: Start 2006-08-18; Study Completion 2015-03-30

CONTACTS AND LOCATIONS:
Overall Officials: Margaret F Keil, C.R.N.P., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Aguila MC, Pickle RL, Yu WH, McCann SM. Roles of somatostatin and growth hormone-releasing factor in ether stress inhibition of growth hormone release. Neuroendocrinology. 1991 Nov;54(5):515-20. doi: 10.1159/000125946. PMID 1684229
- [Background] Albers LH, Johnson DE, Hostetter MK, Iverson S, Miller LC. Health of children adopted from the former Soviet Union and Eastern Europe. Comparison with preadoptive medical records. JAMA. 1997 Sep 17;278(11):922-4. PMID 9302245
- [Background] American Academy of Pediatrics Committee on Early Childhood, Adoption & Dependent Care: Initial medical evaluation of an adopted child. Pediatrics. 1991 Sep;88(3):642-4. No abstract available. PMID 1881750